CLINICAL TRIAL: NCT02025244
Title: Endosonography-Guided Fine-Needle-Aspiration (EUS-FNA) Versus Key Hole Biopsy (KHB) in Diagnostics of Upper Gastrointestinal Submucosal Tumors - a Randomized Trial
Brief Title: EUS-FNA Versus KHB in Diagnostics of Upper Gastrointestinal Submucosal Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Vincent Zoundjiekpon, MD, Vitkovice Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DDC VN 05
Record Dates: First submitted 2012-10-14; First posted 2013-12-31 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Other Specified Disorders of Esophagus, Stomach or Duodenum
Keywords: Key hole biopsy; Upper Gastrointestinal Submucosal Tumors; EUS-FNA; Mitototic Activity; GIST
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Key Hole Biopsy (Active Comparator): Patients with endoscopically detected Upper Gastrointestinal Submucosal Tumors with diameter ≥ 2cm are, according to randomization, allocated to undergo esophagogastroduodenoscopy with Key Hole Biopsy consisting of forceps biopsy through mucosal incision by a needle knife, with subsequent cytological /histological and immunohistochemical evaluation of specimen. In the case of Gastrointestinal Stromal Tumors (GIST), the possibility to determine the mitotic activity is evaluated.
  Interventions: Procedure: Key Hole Biopsy ( KHB); Procedure: EUS-FNA
- EUS-FNA (Active Comparator): Patients with endoscopically detected Upper Gastrointestinal Submucosal Tumors with diameter ≥ 2cm are after randomization allocated to undergo endosonography-guided fine-needle-aspiration biopsy (EUS-FNA) by 22G needle, with subsequent cytological /histological and immunohistochemical examination of the specimen. In the case of Gastrointestinal Stromal Tumors (GIST), the possibility to determine the mitotic activity is evaluated.
  Interventions: Procedure: Key Hole Biopsy ( KHB); Procedure: EUS-FNA

INTERVENTIONS:
Procedure: Key Hole Biopsy ( KHB) — Patients with endoscopically detected Upper Gastrointestinal Submucosal Tumors with diameter ≥ 2cm are, according to randomization, allocated to undergo esophagogastroduodenoscopy with Key Hole Biopsy consisting of forceps biopsy through mucosal incision by a needle knife, with subsequent cytological /histological and immunohistochemical evaluation of specimen. In the case of Gastrointestinal Stromal Tumors (GIST), the possibility to determine the mitotic activity is evaluated.
Procedure: EUS-FNA — Patients with endoscopically detected Upper Gastrointestinal Submucosal Tumors with diameter ≥ 2cm are after randomization allocated to undergo endosonography-guided fine-needle-aspiration biopsy (EUS-FNA) by 22G needle, with subsequent cytological /histological and immunohistochemical examination of the specimen. In the case of Gastrointestinal Stromal Tumors (GIST), the possibility to determine mitotic activity is evaluated. In case of failure of this method, the second one is performed.

SUMMARY:
Upper Gastrointestinal Submucosal Tumors are tumors arising from subepithelial layers of esophageal, gastric or duodenal wall. They usually have an intact mucosa lining on the inner surface. The prognosis and treatment of these tumors depend on their correct diagnostics and mitotic activity in case of Gastrointestinal Stromal Tumors (GIST). A standard forceps biopsy of mucosa is usually not helpful. Therefore, biopsy techniques capable of reaching deeper layer of Upper GUT are needed. The investigators compare KHB and EUS-FNA in the diagnostics of Upper gastrointestinal Submucosal Tumors.

DETAILED DESCRIPTION:
Patients with endoscopically detected submucosal tumors of Upper GUT with diameter ≥ 2cm are enrolled in the trial.

According to randomization, the patients are allocated to either EUS-FNA by 22G needle or KHB consisting of forceps biopsy through mucosal incision by a needle knife, both with subsequent histological/cytological and immunohistochemical evaluation of the specimen. The success of tissue diagnostics was evaluated as well as the possibility to determine the mitotic activity in case of GIST. In case of failure of the initial method, the other method was performed (cross-over design). Patients are hospitalized and kept under observation during 24 hours after the biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Submucosal tumor with endoscopically normal intact mucosa
* Tumor size: 20mm or more
* Localization of tumors: esophagus,stomach, duodenum
* Age: 18 years and older
* The patient´s consent with a diagnostic procedure .

Exclusion Criteria:

* Endoscopically nonbuilding tumor
* Patients younger than 18 years
* Coagulopathy (INR > 1,5, platelets < 100)
* Tumor size < 20mm

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To compare the yield and success of KHB and EUS-FNA in cytological / histological and immunohistochemical diagnostics of Upper Gastrointestinal Submucosal Tumors. | 5 years
  Patients with endoscopically detected Upper Gastrointestinal Submucosal Tumors with diameter ≥ 2cm are randomized and then are allocated to either EUS-FNA by 22G needle or KHB consisting of forceps biopsy through mucosal incision by a needle knife, both with subsequent histological/cytological and imunohistochemical evaluation of the specimen. The success of tissue diagnostics was evaluated.In case of failure of the initial method, the other method was performed (cross-over design).

SECONDARY OUTCOMES:
Detection of mitotic activity in case of Gastrointestinal Stromal Tumors | 5 years
  Patients with endoscopically detected Upper Gastrointestinal Submucosal Tumors with diameter ≥ 2cm are randomized and then allocated to either EUS-FNA by 22G needle or KHB consisting of forceps biopsy through mucosal incision by a needle knife, both with subsequent histological/cytological and imunohistochemical evaluation of the specimen. In case of GIST the possibility to determine the mitotic activity was evalueted.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Zoundjiekpon, MD, Principal Investigator — Vitkovice Hospital
Locations (1):
- Digestive Diseases Center, Vitkovice Hospital, Ostrava, Ostrava, Czechia

REFERENCES:
- [Derived] Zoundjiekpon V, Falt P, Fojtik P, Kundratova E, Mikolajek O, Hanousek M, Reiterova K, Ziak D, Bolek M, Tchibozo A, Kliment M, Urban O. Endosonography-Guided Fine-Needle Aspiration versus "Key-Hole Biopsy" in the diagnostics of upper gastrointestinal subepithelial tumors. A prospective randomized interventional study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2020 Mar;164(1):63-70. doi: 10.5507/bp.2019.013. Epub 2019 Apr 17. PMID 31025658